CLINICAL TRIAL: NCT02895139
Title: Efficacy of Additive Manufactured Orthotic Insoles for the Reduction of Forefoot Plantar Pressure in the Diabetic Foot.
Brief Title: Evaluation of Additive Manufacture in the Production of Orthotic Insoles
Acronym: AMinO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Collaborators: FDM Digital Solutions Ltd (Unknown); East Lancashire Hospitals NHS Trust (Other); Salford Insole (Unknown); Bangor University (Other); iBusiness Flo (Unknown)
Responsible Party: Principal Investigator, Daniel Parker, Principle Investigator, University of Salford
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-1
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes
Keywords: Additive Manufacture; Orthotic Insole
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Additive Manufactured Orthotic Device (Experimental): Device will be produced via additive manufacture to the specification of a Health and Care Professions Council (HCPC) registered orthotist based on a digital foot scan.
  Interventions: Device: Additive Manufactured Orthotic Device
- Moulded Orthotic Device (Other): Historic control collected using same protocol. Intervention was a moulded orthotic device produced from an impression box of the foot shape.
  Interventions: Device: Moulded orthotic
- Milled Orthotic Device (Other): Historic control collected using same protocol. Device will be produced via Computer Aided Design/Computer Aided Manufacture (CAD/CAM) milling to the specification of a HCPC registered orthotist based on a digital foot scan.
  Interventions: Device: Milled orthotic

INTERVENTIONS:
Device: Additive Manufactured Orthotic Device — The 3D foot scan data will be used to generate a 3D model of the foot orthotic which will then be adapted to be suitable for solid printing. The final model will be saved in .stl format for use in the printing software. The additive manufactured orthotic insoles and all features or additions will be produced in a single build from additive materials matched for hardness to medium density EVA. Post production the orthotic will be cleaned to remove support material and a top cover will be attached to the final additive manufactured orthotic insole.
  Arms: Additive Manufactured Orthotic Device
Device: Moulded orthotic — The foam impression box and prescription will be sent to an external company for production of the handmade moulded orthotics. Handmade moulded orthotics will be produced by heating and wrapping medium density Ethylene-vinyl acetate (EVA) around plaster casts of the impression boxes. The orthotic insoles may be manually adapted to meet the requirements of the prescription, this could include cut out sections designed to offload regions of the foot or the addition of features such as metatarsal bars which provide varied support. Features and additions will be added in post manually by cutting and gluing onto the moulded orthotic insole. A top cover will be attached to the final moulded orthotic insole.
  Arms: Moulded Orthotic Device
Device: Milled orthotic — The 3D foot scan data will be used to generate a 3D model of the foot orthotic. This will then be saved in .pan format for use in a CNC milling software. Orthotics and all features will be milled in a single mill from a block of medium density EVA. Post milling the orthotics will be cleaned. The orthotic insoles may be manually adapted to meet the requirements of the prescription, this could include cut out sections designed to offload regions of the foot or the addition of features such as metatarsal bars which provide varied support. Features and additions will be added in post manually by cutting and gluing onto the milled orthotic insole. A top cover will be attached to the final milled orthotic insole.
  Arms: Milled Orthotic Device

SUMMARY:
This study will assess the ability of different orthotic insole treatments to reduce pressure under the ball of the foot. This is important for people who have diabetes because their feet are at higher risk of foot problems in this area. This study will involve the participants wearing a a range of insoles produced by milling, handmade processes and additive manufacture along with normal orthotic footwear. A researcher will measure the pressures under the feet while the participants walk wearing the orthotic insoles.

DETAILED DESCRIPTION:
The study is divided into multiple appointments over which the investigators assess the performance of the orthotic insoles the participants are using.

Screening Appointment (1 hour): The participants will be asked to come to the orthotics department at the Royal Blackburn Hospital. A clinician will perform a routine clinical foot assessment, which will include taking photographs of the feet, to ensure it is safe for the participants to participate in the study. If the participants are not eligible they will not be able to participate in the study, this will not affect the participants normal orthotic care. If the participants are eligible, information on the shape of their feet will be taken using a 3D foot scanner to allow the investigators to produce suitable insoles.

Supply Appointment (1 hour): When the insole is ready the participants will come in for a supply appointment the investigators will check that the insoles and shoes the participants will receive are the correct shape, design and are suitable to wear. At this appointment the investigators will measure the pressure under the feet whilst walking wearing the insoles to check the insole is working correctly. This is done using a thin layer of flexible sensors which go into the participants shoes. The participants will then receive insoles to take home and wear as normal.

After the participants have been supplied with orthotic insoles, a member of the National Health Service (NHS) clinical team will contact them by telephone. This will be each week for the first 4 weeks and then once a month until six months. The call will last no more than 15 minutes and the participants will be asked about their general health, the NHS foot care services they may have used and about the orthotic insoles. In addition at 3 and 6 months after the participants received their orthotic insoles they will be asked to come back into the clinic for a review appointment which will take approximately 1 hour. At these appointments the investigators will measure the pressure under their feet again, using a thin layer of flexible sensors that go into the participants shoes on top of the orthotic insole.

The investigators will also be asking some participants if they would be willing to take part in focus group discussions which will allow more detailed questions to be asked about the participants experiences wearing the orthotic insoles. The participants can decide whether to be involved in these independent of the primary trial. These will be held at the Royal Blackburn Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Are aged between 40 and 85
* Have diabetes
* Have all normal foot structures
* Have sensory neuropathy
* Have detectable pulses in feet
* Have non-standard footwear provided by the orthotics department
* Able to walk 50 meters unaided without stopping

Exclusion Criteria:

* Pregnant or Nursing
* Had prior major injuries to the lower limb (eg. Fractures, skin graft)
* Have active persistent foot or leg ulceration within last 2 years.

The participant may also not be suitable to participate if they have any of the following conditions:

* Ischemia or poor blood supply to your feet
* Charcot Arthropathy
* Connective tissue diseases (for example scleroderma, systemic lupus erythematosus).
* Autoimmune diseases (e.g. rheumatoid arthritis).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Reduction of forefoot pressure to below safety threshold | 6 months
  Number of participants with all forefoot plantar pressure < 200kPa when wearing the orthotic compared to without the orthotic. This will be measured over 6 months of trial to assess if product performance is maintained over duration of use.

SECONDARY OUTCOMES:
Change in forefoot pressure | 6 months
  The affect of the orthotic on forefoot plantar pressure (kPa) at each forefoot site which is above 200kPa without orthotic in participants own footwear. This will be measured over 6 months of trial to assess if product performance is maintained over duration of use.
Patient Outcomes - Quality of Life | 6 months
  Quality of life measure - EuroQol five dimensions questionnaire (EQ-5D)
Patient Outcomes - Capability | 6 months
  Capability and well being measure - ICEpop CAPability measure for Adults (ICECAP-A)
Patient Outcomes - Foot Health | 6 months
  Foot/Pathology status - Foot health status questionnaire.
Patient Outcomes - Orthotic Fit | 6 months
  Percentage of participants own footwear that the orthotics fit into (self-reported %) Compliance (Telephone monitoring)
Organisation outcome - Enquiries | 6 months
  Number of enquiries (e.g. telephone) from patients post dispensing of the orthotics (over 6 months of trial)
Organisation outcome - Appointments | 6 months
  Number of clinical appointments required by patients to address an issue related to the orthotic after fitting. This will be measured over 6 months of trial.
Organisation outcome - Products | 6 months
  Number of footwear products provided by orthotics service. This will be measured over 6 months of trial.
Organisation outcome - Impact on wider healthcare use | 6 months
  Clinical Service Receipt Inventory - primary and secondary health and social care use. This will be measured over 6 months of trial.
Patient Confidence | 6 months
  measured through structured focus group/interviews and narrative analysis: Confidence in products and supply Confidence in prescription and control over design Confidence in colleagues / service provision
Patient experience and satisfaction with orthotics | 6 months
  measured through structured focus group/interviews and narrative analysis: Changes in footwear experiences over 6 months of orthotic use Comfort of orthotics over 6months of orthotic use Satisfaction with orthotics and the service
Patient engagement with health service | 6 months
  measured through structured focus group/interviews and narrative analysis: Need to adjust health behaviour over 6 months of orthotic use Need to seek further assistance for footwear and foot health over 6 months of orthotic use
Clinician confidence in orthotics service | 6 months
  measured through structured focus group/interviews and narrative analysis: Improved evidence base to inform service improvements

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Blackburn Hospital, Blackburn, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No